CLINICAL TRIAL: NCT00489502
Title: Phase I: Clinical Observation of Implementing the MedGem Into a Medical Specialty (i.e. Cardiology) Practice
Brief Title: Clinical Observation of Implementing the MedGem Into a Medical Specialty Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Microlife (Industry)
Other Study IDs: ML002
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Brief Counseling
Device: REE Assessment

SUMMARY:
Due to common CVD diseases associated from obesity, medical providers are in a position to provide assistance. However, less than 10% of all patients receive any weight loss advice from physicians. Perceived barriers to weight loss counseling include lack of self-control of their patients and belief that recommendation is futile, lack of medical training in nutrition, exercise, and obesity management, and lack of insurance reimbursement. Though many barriers are prevalent, research has demonstrated a positive effect with medical advice on the number of obese individuals attempting to lose weight. Analyzing data from the 1996 Behavioral Risk Factor Surveillance System, researchers found, when advised to lose weight by a physician, 78% of overweight patients reported attempting to lose weight. However, if their physician did not discuss weight loss, only 33% of patients within the same BMI category attempted to do so 7. From this information, physicians or allied health staff that provide brief counseling (5-10 minute) along with medical technology that provides basic nutrition assessment might have a positive impact on the number CVD patients that are obese attempting to lose weight.

HYPOTHESIS: Will a medical specialty clinic focused on cardiovascular medicine successfully be able to implement the MedGem device for assessment of basic nutritional needs along with providing "brief" patient education into the medical practice without a house dietitian.

PRIMARY AIMS

1. Can medical staff and/or support staff provide REE assessments (15-minutes) and brief patient education (5-15 minutes) as part of the clinic's operations?
2. Will a third-party payer compensate the Medical Specialty Clinic for the diagnostic procedure CPT Code 94690 for obese patients diagnosed with hypertension (401.1-9, 402.10-11, & 402.90-91), hypercholesterolemia (272.1), and/or hyperlipdemia (272.2)?

SECONDARY AIMS

1. Does self-efficacy increase from REE assessments?
2. Do patients adopt healthy eating (Calorie Reduction and Fat Reduction)following REE assessments?

ELIGIBILITY:
Inclusion Criteria:

* Patients with a BMI (Body Mass Index > 30.0 kg/m2)
* Patients Diagnosed with any of the following ICD-9 Codes: Hypertension (401.1), Hypercholesterolemia (272.1), and/or Hyperlipdemia (272.2-4)
* Patients diagnosed with a secondary ICD-9 Code: Obesity (278) or Morbid Obesity (278.01)

Exclusion Criteria:

* Patients that are pregnant
* Patients under the age of 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-06

CONTACTS AND LOCATIONS:
Overall Officials: Scott McDoniel, M.Ed., Study Director — Microlife USA, Inc.
Locations (1):
- Lake Cardiology, Mt. Dora, Florida, United States